CLINICAL TRIAL: NCT05246618
Title: Phase I FIH Phase I/IIa Randomized Placebocontrolled Doubleblind Trial Evaluating Safety and Tolerability of ExVivo Deceased Donor Kidney Allograft Treatment With TUM012 to Minimize Ischemic Reperfusion Injury After Kidney Transplantation
Brief Title: FIH Phase I/IIa Trial Evaluating Safety of TUM012 to Minimize Ischemic Reperfusion Injury in Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iCoat Medical AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ATMIRe
Record Dates: First submitted 2021-11-28; First posted 2022-02-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Ischemia-reperfusion Injury; Kidney Transplant; Complications
Keywords: Ex-vivo kidney allograft treatment; Transplant outcome
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUM012 (Experimental): Ex-vivo infusion
  Interventions: Drug: TUM012
- Placebo (Placebo Comparator): Ex-vivo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TUM012 — Ex-vivo infusion
  Other Names: Ex-vivo infusion
  Arms: TUM012
Drug: Placebo — Ex-vivo infusion
  Other Names: Ex-vivo infusion
  Arms: Placebo

SUMMARY:
A first-in-human single center, randomized, double-blind, placebo-controlled trial, with primary objective to evaluate safety and tolerability of ex-vivo kidney allograft treatment with TUM012 to reduce ischemia-reperfusion injury in de novo kidney transplant recipients.

DETAILED DESCRIPTION:
Graft ischemia and reperfusion related injury is still the leading cause of graft failure in Deceased Donor kidney transplantation. The aim of the trial is to evaluate the safety of ex-vivo treatment of kidney allografts from deceased-donors with TUM012 to diminish ischemia reperfusion related inflammation, and improve overall transplantat outcome.

ELIGIBILITY:
Inclusion Criteria:

* Standard and extended criteria donor ≥18 years of age, suitable for clinical transplantation and preserved by cold storage.
* Available, personally signed and dated Informed Consent Form (ICF)
* Male or female Chronic Kidney Disease (CKD) patient ≥18 years of age, with Glomerular Filtration Rate (GFR) ≤15 mL/min, awaiting their first kidney transplantation
* ABO-compatible, negative pre-transplant CDC class I and II crossmatch with no Donor Specific Antibodies (DSA), defined as ≤1 000 Mean Fluorescent Intensity (MFI).
* Patient is suitable for surgery, as judged by the investigator
* Completed vaccination program for pneumococcal disease, varicella zoster, measles, and SARS-CoV-2 virus

Exclusion Criteria:

* Surgically induced injuries compromising ex-vivo treatment and/or transplant outcome, as judged by the transplantation surgeon
* Previously undergone any organ and/or cell transplantations
* Patients with positive CDC class I and/or II crossmatch, or negative CDC class I and II crossmatch with pre-existing DSA > 1,000 MFI
* ABO-incompatible DD KT
* Pregnant or breast-feeding woman
* Woman of child-bearing potential, unwilling to use an adequate contraceptive method
* Prior participation in clinical trial with (approved or non-approved) IMP within one month prior to screening for this trial.
* Prior malignancy diagnosis ≤5 years, except for adequately treated basal cell, or squamous cell skin cancer, and cervical carcinoma in situ
* Positive result for serum Human Immunodeficiency Virus (HIV), active hepatitis B-, or C-infection in pre-transplant evaluation
* Clinical signs of ongoing infectious disease, defined as C-Reactive Protein (CRP) >10, unless stable since >4 weeks (<50% increase)
* Concomitant severe conditions requiring treatment and close monitoring, e.g., cardiac failure >grade 3 New York Heart Association (NYHA), unstable coronary disease, or oxygen dependent Chronic Obstructive Pulmonary Disease (COPD)
* History of any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at increased risk because of participation in the trial, or influence the results or the patient's ability to participate in the trial
* Patient unlikely to comply with trial procedures, restrictions, and requirements (e.g., caused by substance abuse, concurrent medical condition, etc.), as judged by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Three months from randomization
  Number of patients with confirmed IMP-related events
Laboratory Analyses (Standard of Care Safety) | Three months from randomization
  Assessment: "normal", "abnormal, not clinically significant", or "abnormal, clinically significant", will as appropriate be reported as Adverse Events.
12-lead Electro-Cardiogram (Standard of Care Safety) | Three months from randomization
  Assessment: "normal", "abnormal, not clinically significant", or "abnormal, clinically significant"
Systolic/diastolic BP (Standard of Care Safety) | Three months from randomization
  Assessment: "normal", "abnormal, not clinically significant", or "abnormal clinically significant"
Pulse Rate (Standard of Care Safety) | Three months from randomization
  Assessment: "normal", "abnormal, not clinically significant", or "abnormal clinically significant"
Peripheral blood oxygenation (Standard of Care Safety) | Three months from randomization
  Assessment: "normal", "abnormal, not clinically significant", or "abnormal clinically significant"
Body temperature (Standard of Care Safety) | Three months from randomization
  Assessment: "normal", "abnormal, not clinically significant", or "abnormal clinically significant"

SECONDARY OUTCOMES:
Exploratory histological evaluation of kidney graft | Three months from randomization
  Biopsy
Exploratory kidney graft function | Three months from randomization
  Number
Exploratory Efficacy: Proteomics | Three months from randomization
  Changed levels from baseline.
Exploratory Efficacy: Markers of IR injury and thromboinflammation plasma level | Three months from randomization
  Changed levels from baseline.
Exploratory Efficacy: Cytokine release plasma level | Three months from randomization
  Changed levels from baseline.
Exploratory Efficacy: Immune cell graft recruitment plasma level | Three months from randomization
  Changed levels from baseline.
Exploratory Efficacy: Pharmacokinetics plasma concentration | Three months from randomization
  Changed levels from baseline.

OTHER OUTCOMES:
Patient survival | One year from randomization
  Number
Incidence of graft rejection | One year from randomization
  Number
Graft survival | One year from randomization
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Ingegerd Dalfelt, Study Director — iCoat Medical AB
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected in this study will be made available to participating trial patients through the investigational site and to the public through publications.
Supporting Information: CSR
Time Frame: After End of Trial
Access Criteria: Individual participant data (IPD) collected in this study will be made available to participating trial patients through the investigational site and to the public through publications, as well as on the company website.
URL: http://www.icoatmedical.com/